CLINICAL TRIAL: NCT00731419
Title: Distal Malignant Biliary Obstruction: A Prospective Randomised Trial Comparing Metal and Plastic Stents in Palliation of Symptomatic Jaundice
Brief Title: Randomised Trial Comparing Metal and Plastic Biliary Stents Stents for Palliating Malignant Jaundice
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cape Town (Other)
Responsible Party: Dr J M Shaw, Department of Surgery, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 144/2007
Record Dates: First submitted 2008-08-05; First posted 2008-08-11 (Estimated); Last update posted 2008-08-11 (Estimated); Status verified 2007-05

CONDITIONS: Biliary Obstruction
Keywords: biliary; obstruction; malignant; stent; palliation
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- SEMS (Active Comparator): Self expanding metal stent compared to plastic stent. Both recognised forms of treatment for condition
  Interventions: Device: SEMS
- Plastic stent (Active Comparator)
  Interventions: Device: SEMS

INTERVENTIONS:
Device: SEMS — Comparing plastic and metal stents
  Other Names: Boston Scientific; biliary self-expanding metal stent; olympus plastic stent

SUMMARY:
Background:

When considering any malignancy with limited life expectancy, palliation and quality of life are paramount. Owing to the limited centres offering ERCP and endoscopic palliation in the South African state sector, patients often travel vast distances and spend large amounts of time away from family and social support structures, severely impairing their quality of life. Stent occlusion with resultant readmission to an ERCP accredited centre obviously compounds this problem.

The hypothesis we propose to test is whether metal stents as a primary procedure result in better patency rates, are more cost effective and improve quality of life than plastic stents. We propose to do this by means of a randomised trial determining the best method of palliation for inoperable distal common bile duct malignancies in the South African context.

Primary end-point Assessing the cost of metal versus plastic stenting in inoperable malignant distal common bile duct strictures in patients with expected survival of 3 months or more as palliation of symptomatic obstructive jaundice. Cost to be assessed in terms of hardware, hospital stay and readmissions for stent occlusion(patency) and complications Secondary end-point Assessing quality of life using a validated scoring system(EORTC QLQ 30) in patients receiving a metal or plastic biliary stent as definitive means of palliation of malignant obstructive jaundice

Hypothesis to be tested Metal stents are superior to plastic stents in terms of patency, resulting in more cost effective palliation of inoperable malignant jaundice and better quality of life due to fewer stent occlusions/episodes of cholangitis.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic jaundice secondary to malignant distal CBD stricture
* Contra-indication to resection (advanced disease/advanced age/poor surgical risk)

Exclusion Criteria:

* Hilar/proximal CBD obstruction
* ECOG performance status 3 or 4
* Duodenal obstruction
* Previous stent placement
* Inability to comply with follow-up
* Ascites and liver metastases
* Not possible to stent endoscopically

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-06; Primary Completion 2009-05 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Overall cost comparison of metal versus plastic stent in patients with limited life expectancy | 6 months

SECONDARY OUTCOMES:
Quality of life assessment | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: John M Shaw, FCS, MMed, Principal Investigator — University of Cape Town
Locations (1):
- Groote Schuur Hospital, Cape Town, Western Cape, South Africa